CLINICAL TRIAL: NCT02672618
Title: Clinical Research to Explore Manifestations of Heart Failure Using Infrared Thermal Imaging Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jing Huang (Other)
Responsible Party: Sponsor-Investigator, Jing Huang, professor，vice director, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: JHuang
Record Dates: First submitted 2016-01-26; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure，Congestive
Keywords: heart failure; infrared thermal imaging
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- chronic heart failure: 18-85years old,having symptoms of heart failure,New York Heart Association（NYHA） class II or above American College of Cardiology/American Heart Association（ACC/AHA） class B, C, including hypertensive heart disease, rheumatic heart disease, ischemic cardiomyopathy and idiopathic cardiomyopathy
- normalCardiac function: 18-85years old,no symptoms of heart failure,NYHA class I or above ACC/AHA class A, including controled hypertension,stability coronary heart disease and rheumatic heart disease
- healthy volunteers: 18-85years old,Without basic cardiovascular diseases

INTERVENTIONS:
Other:  — The IRS system is capable of precisely measuring and storing real-time thermal images with a resolution of 320×240 pixels (IRS S6md Shanghai,China). The camera has Focal Plane Array (FPA), Uncooled microbolometer detector, with a thermal sensitivity of 0.05 ℃ at 20℃ to 30℃. The thermal images were captured at a distance of one meter from the various body regions namely face and the images were analyzed by thermal software（version 1.0）.

SUMMARY:
The purpose of this study is to explore manifestations of Heart Failure Using Infrared Thermal Imaging Technology.

DETAILED DESCRIPTION:
Temperature is a vital and useful indicator for various diseases.Infrared thermal imaging (IRTI) allows the temperature representation of the body surface by thermal distribution, where it depends on the complex relationships defining the heat exchange processes between skin tissue, inner tissue, local vasculature, and metabolic activity.

The decrease in cardiac output in heart failure activate a series of compensatory adaption that are intended to maintain cardiovascular homeostasis. One of most important adaptation is activation of sympathetic nervous system, which could cause peripheral cutaneous vasoconstriction and decrease the skim temperature. Hence, the skim temperature of heart failure would be lower than health people,but which could not discovery by eye. The investigators hypothesize that IRTI could evaluate heart failure by the imaging of temperature distribution in the face on early stages.The aim of this study is to determine the effectiveness of infrared thermal imaging in evaluating heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the trial and sign the informed consent form
2. Aged: 18-85 years
3. Was diagnosed as heart failure
4. There is no trauma, infection, biopsy or puncture, hemorrhage and tumor in the corresponding detection site (face)
5. There is no skin disease, heart, liver, kidney, gastrointestinal tract, hematopoietic system and mental, neurological has no serious diseases

Exclusion Criteria:

1. Fever causes by any reasons, temperature higher than 37.4℃
2. Infection
3. Renal failure
4. Cerebrovascular diseases
5. Moderate anemia or more
6. Not willing to participate in clinical trials

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure patients included in this study had been definitively diagnosed as having with Echocardiography. The healthy volunteer group matched the HF group in number, age, and gender.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Surface temperature (℃）of face and hand measured by Infrared (IR) camera | up to 12 months

SECONDARY OUTCOMES:
LVEF（left ventricular ejection fraction） | up to 12 months
proBNP(pro Brain Natriuretic Peptide) | up to 12 months
catecholamine levels | up to 12 months
Entropy of thermal image | up to 12 months
  Entropy of thermal image: show chaos degree of skim temperature distribution.

CONTACTS AND LOCATIONS:
Overall Officials: hang jing, Study Director — Chongqing Medical University
Locations (4):
- China (4):
  - The 2nd Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - 3Rd People'S Hospital of Chengdu, Chengdu, Sichuan
  - The First Affiliated Hospital of Sichuan Medical University:, Luzhou, Sichuan
  - The First Affiliated Hospital of Chongqing Medical University:, Chongqing

IPD SHARING:
Plan to Share IPD: Yes